CLINICAL TRIAL: NCT02267616
Title: Effectiveness of Prolonged Use of IUD/Implant for Contraception
Acronym: EPIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Susan Thompson Buffett Foundation (Unknown)
Responsible Party: Principal Investigator, Jeffrey Peipert, The Clarence E. Ehrlich Professor; Chair, Dept of Obstetrics and Gynecology, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1603304047
Record Dates: First submitted 2014-10-14; First posted 2014-10-17 (Estimated); Last update posted 2021-04-15 (Actual); Status verified 2021-02

CONDITIONS: Contraception
Keywords: Levonorgestrel intrauterine device (LNG IUD); Etonogestrel (ENG) Implant; Contraception

STUDY DESIGN:
Intervention Model Description: This study will evaluate the use of the Etonogestrel Implant or hormonal intrauterine device (IUD) for contraception past the FDA approved duration. The Etonogestrel Implant is currently approved for 3 years of use, and the hormonal IUD is currently approved for 5 years.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Continued Use Implant Group (Experimental): Woman randomly assigned to the continued use of their Etonogestrel Implant will continue to use their Etonogestrel Implant for contraception past FDA-approved duration of 36 months.
  Interventions: Device: Etonogestrel Implant
- New Implant Group (Active Comparator): Woman randomly assigned to the new Etonogestrel Implant will have their existing Etonogestrel Implant removed and a new implant placed.
  Interventions: Device: Etonogestrel Implant
- Observational Continued Use Group (No Intervention): Women who refuse randomization will have an option of continuing to use their existing Etonogestrel Implant beyond the FDA-approved duration (36 months).

INTERVENTIONS:
Device: Etonogestrel Implant — Subdermal arm implant
  Arms: Continued Use Implant Group; New Implant Group

SUMMARY:
This study will evaluate LNG-IUD and Etonogestrel (ENG) Implant users who are willing to use their contraception beyond the end of the FDA-approved duration. ENG Implant users will also be offered to participate in an arm of the study that will randomize them to either keeping their implant in or having it removed and replaced with a new implant. Participants will be followed for up to three years.

DETAILED DESCRIPTION:
This prospective cohort study will evaluate 675 LNG-IUD users and 675 Etonogestrel (ENG) Implant users who are within 6 months of expiration or beyond the end of the FDA-approved duration. Participants will be contacted via telephone and either scheduled to enroll in person or be mailed the consent form before participation in the EPIC study. After the signed consent form is obtained, participants will also be asked to complete a brief telephone or in-person questionnaire on sociodemographic, medical and reproductive history, sexual and contraceptive history, history of unintended pregnancy and substance abuse. During the informed consent process, implant users will also be offered to participate in an arm of the study that will randomize them (if they consent) to either keeping their subdermal implant in or have it removed and replaced with a new subdermal implant. The randomized control trial subset allows us to compare effectiveness to that of a new implant.

It also allows us to assess "other contraceptive use" (e.g. condom use) in both groups.

Participants will also be asked if they are interested in providing a blood sample for analysis of etonogestrel assay levels at baseline enrollment and annually. If Follow-up phone interviews will occur every 6 months for 36 months beyond the expiration of their method. The investigators will attempt to validate all pregnancy outcomes with medical chart reviews.

ELIGIBILITY:
Inclusion Criteria:

* Women age 18-45
* Within 6 months of expiration or beyond the end of the FDA-approved duration of use of the levonorgestrel intrauterine device (LNG-IUD = 5 years) OR the etonogestrel-releasing subdermal implant (ENG implant = 3 years)
* Able to consent in English or Spanish.
* Not pregnant at the time of enrollment

Exclusion Criteria:

* Have history of female sterilization procedure
* Desire for conception in the next 12 months
* Not sexually active with a male partner

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1076 (Actual)
Dates: Start 2011-12; Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Effectiveness | Three years
  Our primary aim is to test the absolute and relative effectiveness of both the LNG-IUD and the ENG implant in a non-inferiority (equivalence) study comparing failure rates of these methods in the 3 years post-FDA approved duration to the failure rates during the first three years.

SECONDARY OUTCOMES:
Unintended pregnancy rates | Three years
  The contraceptive failure (unintended pregnancy) rates for the LNG-IUD and ENG implant users at 12, 24, and 36 months (after FDA-approved duration of use: 5 years for LNG IUD and 3 years for the ENG implant) of the contraceptive method will be compared to those for CHC users.
Time to contraceptive failure | Three years
  we will use Kaplan-Meier curves to describe the distribution of time to contraceptive failure for the LNG-IUD and ENG implant users compared to combined hormonal contraceptive users (control).
Randomized trial analysis | Three years
  An identical analysis will be performed using the "intention-to-treat" principle (i.e. analyze the participant according to the assigned group as determined by randomization).

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey F Peipert, MD, PhD, Principal Investigator — Indiana University
Locations (2):
- United States (2):
  - Indiana University, Indianapolis, Indiana
  - Washington University in St. Louis School of Medicine, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Henshaw SK. Unintended pregnancy in the United States. Fam Plann Perspect. 1998 Jan-Feb;30(1):24-9, 46. PMID 9494812
- [Background] Singh S, Sedgh G, Hussain R. Unintended pregnancy: worldwide levels, trends, and outcomes. Stud Fam Plann. 2010 Dec;41(4):241-50. doi: 10.1111/j.1728-4465.2010.00250.x. PMID 21465725
- [Background] Goodman S, Hendlish SK, Benedict C, Reeves MF, Pera-Floyd M, Foster-Rosales A. Increasing intrauterine contraception use by reducing barriers to post-abortal and interval insertion. Contraception. 2008 Aug;78(2):136-42. doi: 10.1016/j.contraception.2008.03.008. Epub 2008 Jun 18. PMID 18672115
- [Background] ACOG Committee Opinion no. 450: Increasing use of contraceptive implants and intrauterine devices to reduce unintended pregnancy. Obstet Gynecol. 2009 Dec;114(6):1434-1438. doi: 10.1097/AOG.0b013e3181c6f965. PMID 20134301
- [Background] Peipert JF, Zhao Q, Allsworth JE, Petrosky E, Madden T, Eisenberg D, Secura G. Continuation and satisfaction of reversible contraception. Obstet Gynecol. 2011 May;117(5):1105-1113. doi: 10.1097/AOG.0b013e31821188ad. PMID 21508749
- [Background] Mosher WD, Jones J. Use of contraception in the United States: 1982-2008. Vital Health Stat 23. 2010 Aug;(29):1-44. PMID 20939159
- [Background] Kiriwat O, Patanayindee A, Koetsawang S, Korver T, Bennink HJ. A 4-year pilot study on the efficacy and safety of Implanon, a single-rod hormonal contraceptive implant, in healthy women in Thailand. Eur J Contracept Reprod Health Care. 1998 Jun;3(2):85-91. doi: 10.3109/13625189809051409. PMID 9710712
- [Background] Trussell J. Update on the cost-effectiveness of contraceptives in the United States. Contraception. 2010 Oct;82(4):391. doi: 10.1016/j.contraception.2010.04.008. Epub 2010 May 18. No abstract available. PMID 20851236
- [Background] Trussell J, Lalla AM, Doan QV, Reyes E, Pinto L, Gricar J. Cost effectiveness of contraceptives in the United States. Contraception. 2009 Jan;79(1):5-14. doi: 10.1016/j.contraception.2008.08.003. Epub 2008 Sep 25. PMID 19041435
- [Background] Bahamondes L, Faundes A, Sobreira-Lima B, Lui-Filho JF, Pecci P, Matera S. TCu 380A IUD: a reversible permanent contraceptive method in women over 35 years of age. Contraception. 2005 Nov;72(5):337-41. doi: 10.1016/j.contraception.2004.12.026. Epub 2005 Jul 18. PMID 16246658
- [Background] Makarainen L, van Beek A, Tuomivaara L, Asplund B, Coelingh Bennink H. Ovarian function during the use of a single contraceptive implant: Implanon compared with Norplant. Fertil Steril. 1998 Apr;69(4):714-21. doi: 10.1016/s0015-0282(98)00015-6. PMID 9548163
- [Background] Huber J, Wenzl R. RETRACTED: Pharmacokinetics of Implanon. An integrated analysis. Contraception. 1998 Dec;58(6 Suppl):85S-90S. doi: 10.1016/s0010-7824(98)00120-6. PMID 10095978 (Retraction: PMID 15504385 Rekers H, Affandi B. Contraception. 2004 Nov;70(5):433)
- See also: Institute of Medicine (US). Initial national priorities for comparative effectiveness research. Washington, DC: National Academies Press; 2009. — https://www.google.com/webhp?sourceid=chrome-instant&ion=1&espv=2&ie=UTF-8#q=Initial%20national%20priorities%20for%20comparative%20effectiveness%20research%202009
- See also: Contraceptive technology. 19th rev. ed. New York, N.Y.: Ardent Media; 2007. — http://www.contraceptivetechnology.org/